CLINICAL TRIAL: NCT06732739
Title: Combined Effects of Breathing Teach Back Training And Percussion On Pulmonary Functions In Patients With Pneumonia
Brief Title: Combined Effects of Breathing Teach Back Training And Percussion In Patients With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0370
Record Dates: First submitted 2024-08-13; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia
Keywords: Pneumonia; Percussion; Modified Borg Scale
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percussions with teach-back breathing exercises (Experimental): The treatment will be given with the frequency of 3 times per week for 8 weeks. Treatment sessions will be 25 to 30 minutes with short resting intervals.
  Interventions: Other: percussions with teach-back breathing exercise; Other: PERCUSSION
- percussions (Active Comparator): The treatment will be given with the frequency of 3 times per week for 8 weeks. Treatment sessions will be 25 to 30 minutes with short resting intervals.
  Interventions: Other: PERCUSSION

INTERVENTIONS:
Other: percussions with teach-back breathing exercise — patient will receive Teach Back Breathing Exercises like pursed lip breathing, DE breathing and diaphragmatic breathing Teach-back breathing exercises refer to a method of instructing individuals in breathing techniques and then having them demonstrate or "teach back" the instructions to ensure comprehension and mastery. This educational approach is commonly used in healthcare settings, particularly when teaching patients how to perform various breathing exercises for therapeutic purposes. Patients were informed about the importance of regular chest percussion I will use the clapping technique which provided by cupped hand for 3 minutes in 5 positions of drainage (upper lobes-apical and posterior segment, apical and anterior segment, right upper lobe-posterior segment, left upper lobe-posterior segment, lower lobes- apical segment) with assisted suction three times/shift for four days, and then each patient will be observed.
  Arms: percussions with teach-back breathing exercises
Other: PERCUSSION — similar to Group A, each patient underwent individual interviews. Patients were educated on the significance of regular chest percussion. The clapping technique, executed with cupped hands, was applied for 3 minutes in five drainage positions (upper lobes - apical and posterior segment, apical and anterior segment, right upper lobe - posterior segment, left upper lobe - posterior segment, lower lobes - apical segment). This procedure, including assisted suction three times per shift, was administered for four consecutive days.

SUMMARY:
Pneumonia, marked by lung inflammation, leads to symptoms like fever and difficulty breathing, affecting millions globally. It particularly impacts children and the elderly. Lung function is altered, reducing capacities and obstructing airflow. Post-recovery, patients may experience dyspnea due to lingering fluids-deep breathing exercises, using teach-back training, aid rehabilitation. Combining teach-back with chest percussion in physiotherapy aims to enhance respiratory outcomes in pneumonia patients. This will be a randomized clinical trial sample size calculated by epitool sample size calculator which is 30 patients 15 in each group. Regular chest percussion involves a clapping technique in five drainage positions, with assisted suction. Teach-back breathing exercises will also be implemented in this group In Group A, individuals will perform teach-back breathing exercises with chest percussion. In Group B, a similar protocol will be followed without the teach-back breathing exercises. Data analysis, using SPSS version 21, will include the Shapiro-Wilk Test for normality assessment. Descriptive statistics, paired sample t-tests, Wilcoxon signed-rank tests, independent sample t-tests, and Mann-Whitney U tests will be employed to analyze group measurements, changes over time, and differences between groups. This comprehensive approach aims to provide a thorough understanding of the study variables and measurements.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 35-45 years
* Diagnosed pneumonia

Exclusion Criteria:

* History of neurological disorders
* History of fractures
* History of other pulmonary complications (15)
* Patients having any chest infection will be excluded

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary functions test | baseline and fourth week
  A pulmonary function test (PFT) is a diagnostic assessment that evaluates the functional capacity of the respiratory system, providing valuable information about lung volumes, capacities, and the efficiency of gas exchange. These tests are crucial for diagnosing and monitoring respiratory conditions such as asthma, chronic obstructive pulmonary disease , and restrictive lung diseases, Pulmonary function test Normal values are FEV1 80% to 120%, FVC 80% to 120%. Absolute FEV1 /FVC ratio, Within 5% of the predicted ratio, TLC 80% to 120%
SF 36 | baseline and fourth week
  The SF-36, or Short Form 36, is a widely used questionnaire designed to assess an individual's health-related quality of life. It encompasses 36 questions across eight health domains, providing insights into various aspects of physical and mental well-being. The questionnaire covers areas such as physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Social Security Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris AM, Huang L, Bacchetti P, Turner J, Hopewell PC, Wallace JM, Kvale PA, Rosen MJ, Glassroth J, Reichman LB, Stansell JD. Permanent declines in pulmonary function following pneumonia in human immunodeficiency virus-infected persons. The Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):612-6. doi: 10.1164/ajrccm.162.2.9912058. PMID 10934095
- [Background] Rudan I, Tomaskovic L, Boschi-Pinto C, Campbell H; WHO Child Health Epidemiology Reference Group. Global estimate of the incidence of clinical pneumonia among children under five years of age. Bull World Health Organ. 2004 Dec;82(12):895-903. Epub 2005 Jan 5. PMID 15654403
- [Background] Hogan DR, Stevens GA, Hosseinpoor AR, Boerma T. Monitoring universal health coverage within the Sustainable Development Goals: development and baseline data for an index of essential health services. Lancet Glob Health. 2018 Feb;6(2):e152-e168. doi: 10.1016/S2214-109X(17)30472-2. Epub 2017 Dec 13. PMID 29248365